CLINICAL TRIAL: NCT04507282
Title: Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi
Brief Title: Eosinophil and Anticoagulation in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Bursa Postgraduate Hospital (Other)
Responsible Party: Principal Investigator, Hasan ARI, Medical Doctor of Cardiology, Bursa Postgraduate Hospital
Other Study IDs: Bursa Postgraduate Hospital
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COVID 19 positive patients
  Interventions: Drug: LMWH

INTERVENTIONS:
Drug: LMWH — COVID 19 positive patients anticogulation level, subprophylactic level and prophylactic level

SUMMARY:
Despite prophylactic anticoagulant treatments, thrombotic complications may develop in patients with Coronavirus disease 2019 (COVID-19). This study aimed to evaluate anti-Factor Xa levels to determine the anticoagulant activity of low molecular weight heparin (LMWH) in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years, who were diagnosed with COVID-19 and were administered LMWH,
* agreed to participate in the study were included

Exclusion Criteria:

* Patients with previous coagulopathy,
* continuous indication of anticoagulant therapy (atrial fibrillation (AF), valve disease),
* glomerular filtration rate (GFR) <30 mL/min or undergoing dialysis, or with known liver dysfunction were excluded from the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID 19 positive patients treated with LMWH
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
subprophylactic anticogulation level | 14 days
  <0.2IU/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yüksek İhtisas Hastanesi, Yıldırım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ari S, Can V, Demir OF, Ari H, Agca FV, Melek M, Camci S, Dikis OS, Huysal K, Turk T. Elevated eosinophil count is related with lower anti-factor Xa activity in COVID-19 patients. J Hematop. 2020 Oct 8;13(4):249-258. doi: 10.1007/s12308-020-00419-3. eCollection 2020 Dec. PMID 33046998